CLINICAL TRIAL: NCT05618821
Title: Clinical Outcomes of Indocyanine Green Tracer Using in Laparoscopic Gastrectomy With Lymph Node Dissection for Remnant Gastric Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fujian Medical University (Other)
Responsible Party: Principal Investigator, Chang-Ming Huang, Prof., Professor, Fujian Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FUGES-027
Record Dates: First submitted 2022-06-03; First posted 2022-11-16 (Actual); Last update posted 2022-11-16 (Actual); Status verified 2022-11

CONDITIONS: Gastric Cancer
Keywords: Indocyanine Green Tracer; Laparoscopic Gastrectomy; Remnant Gastric Cancer
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ICG (Experimental): Laparoscopic gastrectomy Group with the use of near-infrared imaging (ICG group)
  Interventions: Drug: Indocyanine Green Tracer
- Non-ICG (Active Comparator): Laparoscopic gastrectomy Group without the use of near-infrared imaging (Non-ICG group)
  Interventions: Drug: Indocyanine Green Tracer

INTERVENTIONS:
Drug: Indocyanine Green Tracer — Laparoscopic gastrectomy with lymph node dissection for remnant gastric cancer using Indocyanine Green Tracer

SUMMARY:
Patients with resectable remnant gastric cancer were selected as study subjects to investigate the safety, efficacy, and feasibility of ICG near-infrared imaging tracing in guiding laparoscopic lymph node dissection for remnant gastric cancer by comparing injection ICG group and non-injection ICG group.

DETAILED DESCRIPTION:
Indocyanine Green Tracer is often applied in surgery for gastric cancer. Its application in laparoscopic gastrectomy with lymph node dissection for remnant gastric cancer is at the stage of cases accumulation, method studying and clinical research. There is no prospective studies to identify the clinical outcomes of Indocyanine Green Tracer using in laparoscopic gastrectomy with lymph node dissection for remnant gastric cancer. On the basis of more than 300 cases of laparoscopic gastrectomy with lymph node dissection for remnant gastric cancer, we want to apply the Indocyanine Green Tracer, a cheap, easy to operate and no radiation pollution way, to predict the positive lymph nodes in remnant gastric cancer, to guid the scope of laparoscopic lymph node dissection for remnant gastric cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Age from 18 to 75 years
2. Remnant gastric cancer (cT1-4a, N-/+, M0 at preoperative evaluation according to the American Joint Committee on Cancer (AJCC) Cancer Staging Manual Seventh Edition)

(4) No distant metastasis, no direct invasion of pancreas, spleen or other organs nearby in the preoperative examinations (5) Performance status of 0 or 1 on the ECOG (Eastern Cooperative Oncology Group) scale (6) ASA (American Society of Anesthesiology) class I to III (7) Written informed consent

Exclusion Criteria:

1. Women during pregnancy or breast-feeding
2. Severe mental disorder
3. History of previous upper abdominal surgery (except for laparoscopic cholecystectomy and gastrectomy)
4. History of previous gastric surgery (including ESD/EMR for gastric cancer)
5. Rejection of laparoscopic resection
6. History of allergy to iodine agents
7. Enlarged or bulky regional lymph node diameter over 3cm by preoperative imaging
8. History of other malignant disease within past five years
9. History of previous neoadjuvant chemotherapy or radiotherapy
10. History of unstable angina or myocardial infarction within the past six months
11. History of unstable angina or myocardial infarction within past six months
12. History of continuous systematic administration of corticosteroids within one month
13. Requirement of simultaneous surgery for another disease
14. Emergency surgery due to complications (bleeding, obstruction or perforation) caused by gastric cancer
15. FEV1<50% of the predicted values
16. Linitis plastica, Widespread

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Estimated)
Dates: Start 2022-06-03 (Actual); Primary Completion 2025-04-01 (Estimated); Study Completion 2028-04-01 (Estimated)

PRIMARY OUTCOMES:
Total Number of Retrieved Lymph Nodes | 30 days
  Total Number of Retrieved Lymph Nodes

SECONDARY OUTCOMES:
Lymph node noncompliance rate | 30 days
  Lymph node noncompliance rate
Relationship between fluorescent lymph nodes in the ICG group and total number of lymph nodes in the ICG group | 30 days
  Relationship between fluorescent lymph nodes in the ICG group and total number of lymph nodes in the ICG group
Relationship between fluorescent lymph nodes in the ICG group and positive lymph nodes in the ICG group (positive rate) | 30 days
  Relationship between fluorescent lymph nodes in the ICG group and positive lymph nodes in the ICG group (positive rate)
Relationship between fluorescent lymph nodes in the ICG group and negative lymph nodes in the ICG group (false positive rate) | 30 days
  Relationship between fluorescent lymph nodes in the ICG group and negative lymph nodes in the ICG group (false positive rate)
Relationship between non-fluorescent lymph nodes in the ICG group and negative lymph nodes in the ICG group (negative rate) | 30 days
  Relationship between non-fluorescent lymph nodes in the ICG group and negative lymph nodes in the ICG group (negative rate)
Number of Metastasis Lymph Nodes | 30 days
  Number of Metastasis Lymph Nodes
Metastasis rate of lymph node | 30 days
  Metastasis rate of lymph node
Postoperative morbidity rate | 30 days
  Postoperative morbidity rate
Postoperative mortality rate | 30 days
  Postoperative mortality rate
3-year overall survival rate | 3 years
  3-year overall survival rate
3-year disease-free survival rate | 3 years
  3-year disease-free survival rate
3-year recurrence pattern | 3 years
  3-year recurrence pattern
Postoperative recovery course | 30 days
  Time to first ambulation, flatus, liquid diet and soft diet, and postoperative hospital stay
Intraoperative situation | 30 days
  Operation time, intraoperative blood loss, and intraoperative morbidity rate

CONTACTS AND LOCATIONS:
Locations (1):
- Fujian Medical University Union Hospital, Fuzhou, Fujian, China

IPD SHARING:
Plan to Share IPD: Undecided